CLINICAL TRIAL: NCT04791969
Title: The ION+EMI Study: Intermittent Oral Naltrexone Enhanced With an Ecological Momentary Intervention for Methamphetamine-using MSM
Brief Title: Intermittent Oral Naltrexone Enhanced With an Ecological Momentary Intervention for Methamphetamine-using MSM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glenn-Milo Santos (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Glenn-Milo Santos, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-32912; R01DA053171 (NIH)
Record Dates: First submitted 2021-01-19; First posted 2021-03-10 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Methamphetamine Use Disorder
Keywords: Methamphetamine; meth; naltrexone
MeSH Terms: interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: 2:1 Naltrexone with EMI vs. Placebo with EMI
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind, placebo controlled 2b clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naltrexone with ecological momentary intervention (Experimental): Naltrexone Hydrochloride, 50 mg., intermittent with ecological momentary assessment (EMA)
  Interventions: Drug: Naltrexone Hydrochloride; Behavioral: Ecological Momentary Intervention
- Placebo with ecological momentary intervention (Placebo Comparator): Placebo, intermittent with ecological momentary assessment (EMA)
  Interventions: Drug: Placebo; Behavioral: Ecological Momentary Intervention

INTERVENTIONS:
Drug: Naltrexone Hydrochloride — Intermittent Oral Naltrexone, 50 mg
  Other Names: ReVia
  Arms: Naltrexone with ecological momentary intervention
Drug: Placebo — Intermittent Oral Placebo
  Arms: Placebo with ecological momentary intervention
Behavioral: Ecological Momentary Intervention — Receive ecological momentary intervention if ecological momentary assessment reports meth craving, stress, not taking study drug, or antecedents detected for "high risk" meth use.
  Other Names: EMI

SUMMARY:
This is a double-blind, placebo-controlled phase 2b trial in which 54 MSM who use meth will be randomly assigned (2:1) to receive 12 weeks of as-needed intermittent oral naltrexone 50 mg enhanced with an EMA-informed EMI platform, or receive as-needed placebo with EMA-informed EMI. The 12-week treatment period is consistent with other pharmacotherapy trials for substance use disorders. The proposed sample size is also consistent with other phase 2b trials for substance use treatment. Upon enrollment, participants will complete daily EMA assessments and weekly visits for behavioral surveys and urine testing for meth metabolites, study drug dispensing and computer-based counseling for substance use. Safety laboratory assessments and vital signs will be completed monthly. Efficacy (Specific Aims 1-3) will be assessed upon trial completion as measured by proportion meth-positive urine samples; PrEP and ART adherence by drug levels and viral load testing; and sexual risk behavior data accounting for PrEP use and viral suppression.

DETAILED DESCRIPTION:
Methamphetamine (meth) use is very common among men who have sex with men (MSM), particularly MSM living with HIV. Meth use among HIV-negative and HIV-positive MSM is up to 13 and 34 times more prevalent than in the general U.S. adult population, respectively. Meth use is independently associated with HIV-related sexual risk behaviors among MSM and can function as a barrier to antiretroviral therapy (ART) and pre-exposure prophylaxis (PrEP) adherence. Thus, effective interventions to reduce meth use may also function as an important HIV prevention and care intervention by reducing meth-related HIV risk behavior, and optimizing ART and PrEP adherence. MSM comprise two-thirds of the new infections in the United States. Despite this continued domestic HIV epidemic and the high prevalence of meth use among MSM, few interventions have proven efficacious for MSM who use meth. The investigators seek to address this gap by evaluating the efficacy of intermittent oral naltrexone enhanced with an ecological momentary intervention (ION+EMI) for meth use treatment. Naltrexone, a µ-opioid receptor antagonist, is a promising agent for MSM who use meth. Meth is rapidly metabolized to amphetamine in the bloodstream and daily naltrexone has shown efficacy in reducing amphetamine urine-positivity and relapse. Oral naltrexone is inexpensive and has few toxicities, but the standard daily regimen for naltrexone hampers compliance as patients frequently neglect to take the medication. Alternate regimen schedules have been proposed to increase efficacy and expand the population that may benefit from this pharmacologic agent. One alternative approach is the targeted administration of intermittent oral naltrexone (ION), whereby individuals are instructed to take the medication as needed in anticipation of substance use, after exposure to triggers of substance use, or during periods of craving. Administration of naltrexone prior to exposure to amphetamines significantly attenuated amphetamine craving in 4 trials. Additionally, emerging evidence suggests that ecological momentary interventions (EMI) that respond to in-the-moment contexts can lead to positive health behaviors, such as increasing medication dosing. EMI are particularly well-suited to enhancing as-needed dosing of naltrexone because anticipation of meth use and meth craving in a natural setting changes within a person from moment to moment, and the detection of these momentary fluctuations can support the delivery of just-in-time messages to encourage medication use to prevent participants from proceeding from craving to meth use. A pilot study led by our research team on ION found that meth-using MSM who use at least 1 day per week had significantly greater reductions in meth-using days when treated with as-needed naltrexone, compared to placebo. Moreover, naltrexone participants had greater reductions in serodiscordant receptive anal intercourse and serodiscordant condomless receptive anal intercourse, compared to placebo. In the pilot, participants reported taking study drug 64% of the days that they craved or anticipated meth use. Participants also completed ecological momentary assessments (EMA) with a 74% response rate, indicating that real-time assessments are feasible and acceptable. To build on the results of this study and 4 other naltrexone trials, the investigators propose to evaluate intermittent naltrexone to treat meth in a phase 2b efficacy trial supplemented by an EMA-informed EMI that responds to a participant's real-time craving levels or anticipated meth use to provide in-the-moment medication reminders when participants would most benefit from naltrexone. The investigators hypothesize that pairing ION with EMI will further amplify reductions in meth use by providing just-in-time reminders for naltrexone to optimize adherence, thereby interrupting the progression from craving to meth use.

ELIGIBILITY:
Inclusion Criteria:

* cisgender male (male gender and sex assigned at birth)
* age 18-70 years* (naltrexone's tolerability and safety has been demonstrated among older adults up to age 70)
* self-reported condomless anal sex with men or missing Pre-Exposure Prophylaxis or antiretroviral therapy doses due to meth use in the prior three months while under the influence of meth
* self-reported meth use at least weekly
* mild, moderate or severe meth use disorder
* positive meth sample via sweat patch or urine testing during screening
* interested in reducing meth use
* no current acute illness requiring prolonged medical care
* no chronic illness that is likely to progress clinically during trial
* able and willing to provide informed consent and adhere to visit schedule
* current CD4 count ≥ 200 cells/mm3; or CD4 count of 100-199 cells/mm3 and HIV viral load < 200 copies/mL (if living with HIV)
* baseline complete blood count, total protein, albumin, glucose, alkaline phosphatase, creatinine, blood urea nitrogen test, and electrolytes without clinically significant abnormalities as determined by study clinician in conjunction with symptoms, physical exam, and medical history

Exclusion Criteria:

* any psychiatric (e.g., depression with suicidal ideation) or medical condition that would preclude safe participation
* known allergy or prior adverse reaction to naltrexone
* current use of any opioids or a known medical condition which currently requires or may likely require opioid analgesics
* opioid-positive urine test at screen/enrollment visits (naltrexone can induce opioid withdrawal)
* moderate or severe liver disease (aspartate aminotransferase test, alanine aminotransferase test, or total bilirubin > 3 times upper limit of normal)
* impaired renal function (creatinine clearance < 60 ml/min)
* currently participating in another intervention research study with potential overlap
* severe alcohol use disorder as determined by structured clinical interview for DSM-5 criteria
* any condition that, in the PI and/or study clinician's judgment interferes with safe participation or adherence to study procedures

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cisgender male, men who have sex with men
Enrollment: 60 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn-Milo Santos, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Department of Public Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Additional participants were enrolled to account for higher than anticipated lost to follow-up during study. Enrollment sample approved by funder (National Institutes of Health), study Institutional Review Board and study data safety monitoring board.
Period: Overall Study
Arm/Group | Naltrexone With Ecological Momentary Intervention | Placebo With Ecological Momentary Intervention
Started | 40 | 20
Completed | 35 | 11
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone With Ecological Momentary Intervention | Placebo With Ecological Momentary Intervention | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.58 (13.51) | 44.65 (7.79) | 43.93 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 39 | 20 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 3 | 14
  Not Hispanic or Latino | 29 | 17 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 20 | 14 | 34
  More than one race | 7 | 0 | 7
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 40 | 20 | 60
Number of meth-using Male Partners [Mean (Standard Deviation); unit: number of meth-using male partners] | 2.03 (1.29) | 2.3 (1.08) | 2.12 (1.22)
Meth positive urine sample [Count of Participants; unit: Participants] | 35 | 18 | 53
PrEP drug levels detected (PrEP Adherent) or Virally Suppressed (Antiretroviral treatment adherent) [Count of Participants; unit: Participants] | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of People With Meth-positive Urine Tests at Weekly Visits
Description: As measured by the count of participants with meth-positive urine tests.
Time Frame: Every week from week 1 to the end of treatment at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone With Ecological Momentary Intervention | Placebo With Ecological Momentary Intervention
Number analyzed (Participants) | 40 | 20
Participants
  Week 1 | 20 | 13
  Week 2 | 23 | 9
  Week 3 | 21 | 10
  Week 4 | 25 | 10
  Week 5 | 19 | 8
  Week 6 | 16 | 8
  Week 7 | 19 | 7
  Week 8 | 19 | 5
  Week 9 | 17 | 9
  Week 10 | 19 | 9
  Week 11 | 23 | 9
  Week 12 | 27 | 9

2. Secondary Outcome: Mean in Sexual Risk Behaviors at Week 12
Description: As measured by the mean number of sexual partners with whom they used meth, in the prior month, at week 12
Time Frame: Past month behavior, measured at the end of treatment at 12 weeks
Population: Participants who completed sexual behavior questionnaire at final visit
Measure: Mean (Standard Deviation); unit: number of meth-using male partners
Arm/Group | Naltrexone With Ecological Momentary Intervention | Placebo With Ecological Momentary Intervention
Number analyzed (Participants) | 35 | 11
number of meth-using male partners | 1.23 (1.19) | 1.0 (1.10)

3. Other Pre Specified Outcome: Adherent to PrEP or to Antiretroviral Medication
Description: As measured by PrEP drug levels being detected in HIV negative participants (PrEP Adherent and viral suppression rates in HIV positive participants (Antiretroviral treatment adherent)
Time Frame: At the end of treatment at the 12-week visit
Population: Participants who are HIV-negative and who provided samples for PrEP drug levels testing at final visit, or participants who are living with HIV and provided samples for HIV viral load testing
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone With Ecological Momentary Intervention | Placebo With Ecological Momentary Intervention
Number analyzed (Participants) | 21 | 9
Participants | 15 | 7

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events are assessed weekly by study clinician and also through the monthly safety lab tests
Arm/Group | Naltrexone With Ecological Momentary Intervention | Placebo With Ecological Momentary Intervention
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/40 | 0/20
Other Adverse Events (participants affected / at risk) | 7/40 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone With Ecological Momentary Intervention (N=40) | Placebo With Ecological Momentary Intervention (N=20)
Post-obstructive renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) — Post-obstructive renal failure led to in patient hospitalization
Hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Hernia present since 2017, but resulted in hospitalization on 3/20/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone With Ecological Momentary Intervention (N=40) | Placebo With Ecological Momentary Intervention (N=20)
Fatigue (General disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations include loss to follow-up in study participants, leading to a smaller number of observations analyzed than original number of participants enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT04791969/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT04791969/SAP_001.pdf